CLINICAL TRIAL: NCT06218225
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effects of an Immune-boosting Food Supplement on the Severity and Frequency of Pediatric Respiratory Tract Infections
Brief Title: Effect of an Immune-boosting Food Supplement on the Severity and Frequency of Pediatric Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMMUNOJR
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-11

CONDITIONS: Immunomodulation; Respiratory Tract; Infection, Upper (Acute)
MeSH Terms: conditions — Infections | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: Randomized double blind verum vs placebo
Who Masked: Participant, Care Provider
Masking Description: Different batch code assigned to products, same labeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Partecipants received a food supplement with the innovative IMMUREMEDY®-B complex and Lactobacillus rhamnosus CRL1505.
  Interventions: Dietary Supplement: Verum
- Placebo (Placebo Comparator): Partecipants received a food supplement in the same primary packaging of the verum, but without active substances
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Verum — 1st cycle - 30 days continuous use Cycle 2 - first 15 days washout, remaining 15 days use of study product Cycle 3 - first 15 days washout, remaining 15 days use of study product 4th cycle - 30-day washout
  Arms: Verum
Dietary Supplement: Placebo — 1st cycle - 30 days continuous use Cycle 2 - first 15 days washout, remaining 15 days use of placebo Cycle 3 - first 15 days washout, remaining 15 days use of placebo 4th cycle - 30-day washout
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of the product in developing immune reinforcement that results in decreased susceptibility to respiratory infections of viral origin in children aged 3 to 10 years with a number of respiratory tract infectious events in the previous year greater than 4. The main questions it aims to answer are:

* Has the number of infectious events been reduced from last year?
* Does the severity of symptoms decrease with the use of the product?

Participants will be treated for 4 months. Treatment efficacy will be evaluated by:

* 2 scheduled visits with the investigating pediatrician (T0 - enrollment and start of treatment; T1- end of treatment).
* Verification of progress during the study by scheduled telephone meetings.
* The use of a diary where the patient or parent/caregiver will report all events (even mild) affecting the respiratory tract, taking care to fully complete the Wisconsin Upper Respiratory Symptom Survey for kids (WURSS-k) questionnaire.

DETAILED DESCRIPTION:
The immune system is a complex network consisting of organs, tissues, cells and the substances they produce. It has the function of protecting the body from external agents (including infectious agents) by activating three different types of response: the innate response, the adaptive response, and the mechanical or chemical response. The innate and adaptive response are activated together, one modulating the other. The innate or natural response represents a first line of defense. The adaptive or specific response is a slower but more powerful and targeted defensive response and enables the creation of immunological memory.

In the pediatric setting in the early months, and in the later first years of life, where the "immunological memory" has not yet strengthened, infectious events such as fever, flu, colds, throat discomfort, cough, respiratory infections, sore throat, various respiratory tract ailments, gastrointestinal diseases or related only to the intestinal tract occur frequently. It will take time for it to strengthen, and for the little one to be immune to a bacterial infection, but there are remedies to help. A healthy lifestyle, physical activity and a balanced diet that allows the right amount of protein, vitamins and minerals can strengthen the immune system. In some cases, where healthy diet and lifestyle needed support, the use of natural substances with immune-stimulating action proves useful.

The tested product is a dietary supplement specifically designed to modulate immune defenses in children. It contains the innovative IMMUREMEDY®-B complex and Lactobacillus rhamnosus CRL1505. Zinc and vitamins B6, B12, C, and D contribute to normal immune system function. Elderberry and acerola support the body's natural defenses. Lactobacillus rhamnosus CRL1505 is a probiotic that promotes the balance of the flora intestinal flora. Several clinical studies have shown that it can reduce the incidence of pediatric infections, including respiratory tract infections.

The goal of this clinical trial is to evaluate the efficacy of the product in developing immune reinforcement that results in decreased susceptibility to respiratory infections of viral origin in children aged 3 to 10 years with a number of respiratory tract infectious events in the previous year greater than 4.

Treatment consists of taking one single-dose bottle daily for a total of 4 months as follows:

1st cycle - 30 days use of study product or placebo Cycle 2 - first 15 days washout, remaining 15 days use of study product or placebo Cycle 3 - first 15 days washout, remaining 15 days use of study product or placebo 4th cycle - 30-day washout Numerosity and severity of infectious events will be assessed during meetings with the pediatrician and through a diary where the patient or parent/caregiver will report all events (even mild) affecting the respiratory tract, taking care to fully complete the Wisconsin Upper Respiratory Symptom Survey for kids (WURSS-k) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes children aged 3-10 years, with a number of respiratory tract infectious events in the previous year greater than 4.

Exclusion Criteria:

* Acute upper respiratory tract or other infection within 7 days prior to enrollment, cystic fibrosis, immunodeficiency syndromes, abnormalities respiratory tract anatomy, use of immunostimulant drugs or immunosuppressants in the previous 4 weeks.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the reduction in the severity of symptoms related to Acute Respiratory Tract Infections | For each infectious event, it should be filled in on the first day of symptoms, on the third day of symptoms, and if symptoms persist, it should also be filled in on the seventh day of symptoms.
  Evaluation of the reduction of illness-specific symptoms during an ARI by means of validated 15-items questionnaire (WURSS-k)

SECONDARY OUTCOMES:
Evaluation of the reduction in the number of Acute Respiratory Tract Infections | T0 (first visit), T1 (4 months later - end of treatment)
  Evaluation of the reduction in the number of infectious events during the 4-months study duration, based on how many times each patient completed the WURSS-k questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Gioacchino Calapai, Messina, Italy